CLINICAL TRIAL: NCT04814914
Title: An Observational Study to Evaluate the Presence of Symptoms After COVID-19 Infection in Patients Who Participated in K031-120 or K032-120 Study ("Long Hauler")
Brief Title: An Observational Clinical Study to Evaluate COVID-19 Symptoms in "Long Hauler" Patients Who Participated in K031-120 or K032-120
Status: Completed | Type: Observational
Sponsor: Kaleido Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: K034-120
Record Dates: First submitted 2021-03-23; First posted 2021-03-24 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
Keywords: Microbiome; COVID-19; Corona Virus; Corona Virus Disease; Kaleido; Kaleido Biosciences; KB109; Oligosaccharide; Glycan; Microbiome metabolic therapy; MMT; Supportive Self Care; SSC; Telemedicine; K031-120; K032-120
MeSH Terms: conditions — COVID-19 | interventions — Single Person

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- KB109 + Self Supportive Care (SSC)
  Interventions: Other: KB109 + Self Supportive Care
- Self Supportive Care (SSC) Alone
  Interventions: Other: Self Supportive Care (SSC) Alone

INTERVENTIONS:
Other: KB109 + Self Supportive Care — KB109 is a novel glycan
  Groups: KB109 + Self Supportive Care (SSC)
Other: Self Supportive Care (SSC) Alone — Self Supportive Care (SSC) Alone
  Groups: Self Supportive Care (SSC) Alone

SUMMARY:
This observational clinical study aims to evaluate the presence of symptoms of COVID-19 infection in patients who participated in K031-120 or K032-120 ("long hauler").

ELIGIBILITY:
Inclusion Criteria:

* Have consented to participate over the telephone
* Have been randomized in either the K031-120 or K032-120 study

Exclusion Criteria:

* Have withdrawn consent from K031-120 or K032-120

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who participated in K031-120 or K032-120 study.
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with persistent COVID-19 symptoms for at least 12-weeks post-randomization in K031-120 or K032-120 study. | 12-weeks from randomization in K031-120 or K032-120

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wingertzahn, PhD, Study Director — Kaleido Biosciences, Inc.
Locations (2):
- United States (2):
  - HealthStar Research, LLC, Hot Springs, Arkansas
  - Quad Clinical Research, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No